CLINICAL TRIAL: NCT02489201
Title: A Phase 1B Study of Donafenib Monotherapy in Advanced Oesophageal Cancer Progressing After Chemotherapy
Brief Title: A Study of Donafenib Monotherapy in Advanced Oesophageal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Corporate policy adjustments
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZGDE1B
Record Dates: First submitted 2015-06-24; First posted 2015-07-02 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Oesophageal Cancer
Keywords: donafenib
MeSH Terms: conditions — Esophageal Neoplasms | interventions — donafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- donafenib tosilate tablets (Experimental): 200mg bid
  Interventions: Drug: donafenib tosilate tablets

INTERVENTIONS:
Drug: donafenib tosilate tablets — 200mg,bid
  Other Names: CM4307

SUMMARY:
This open-label, one-center, noncomparative, two-stages phase 1B trial assessed the tyrosine kinase inhibitor donafenib tosylate tablets(400 mg/d,200mg bid) in patients with advanced, inoperable oesophageal cancer progressing after chemotherapy .

The primary endpoint is the safety.The secondary endpoints are tumor response and progression-free survival.

DETAILED DESCRIPTION:
This open-label, noncomparative, two-part phase 1B trial recruited patients with advanced, inoperable oesophageal cancer. The primary objectives were to assess the safety for donafenib tosylate tablets .The secondary objectives were to estimate tumor response, progression-free survival, duration of response, and disease control rate (response plus stable disease); to evaluate changes in quality of life(QoL); This study is 2-stages designing. The investigators plan to enroll 19 patients in the first stage study. The investigators will start the secondary stage study if the disease control rate >=8/19.

ELIGIBILITY:
Inclusion Criteria:

* All patients provided written, informed consent.
* Have histologically confirmed advanced oesophageal squamous-cell carcinoma, or type I/II Siewert junctional tumours.
* Have received up to two previous chemotherapy regimens( Platinum containing regimens & Paclitaxel / docetaxel containing regimens).
* Have an Eastern Cooperative Oncology Group Performance status of 0-1.
* Have ability to swallow tablets.
* no contraindications to sorafenib or donafenib.
* Have either measurable or evaluable lesion on CT.

Exclusion Criteria:

* Patients with brain metastases.
* Patients receiving cytotoxic chemotherapy, immunotherapy or hormonal therapy, radiotherapy to site of measurable or evaluable disease within the previous 4 weeks.
* Patients had evidence of clinically active interstitial lung disease or abnormal blood results by predefined criteria (serum bilirubin >1.5 times upper limit of reference range, aspartate or alanine aminotransferase>2.5 times the upper limit of normal if no demonstrable liver disease) .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | 54 weeks
  percentage of any adverse events

SECONDARY OUTCOMES:
Tumor response | 54 weeks
  Tumor evaluation by investigators according to RECIST 1.1 criteria
Progression-free survival | 54 weeks
  PFS was defined as the time from date of randomization to disease progression radiological or death due to any cause, whichever occurs first. Subjects without progression or death at the time of analysis were censored at their last date of tumor evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Xu, Doctor, Principal Investigator — The Affiliated Hospital of Military Medical Science
Locations (1):
- Affiliated Cancer Center of Academy of Military Medical Sciences, Beijing, China